CLINICAL TRIAL: NCT04701723
Title: Interest of Cardiac Coherence in the Prevention of Chronic Post-traumatic Stress Disorder: Pilot Study
Acronym: COHEPS-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019/CHU/02
Record Dates: First submitted 2020-12-23; First posted 2021-01-08 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Coherence Training (Experimental): The cardiac coherence training will consist in the realization during 3 months by the patient, at home :
  * of 6 respiratory cycles by minute (inspiration : 4,5 seconds/expiration : 5,5 seconds),
  * during 5 minutes,
  * 3 times a day (morning, late morning and late afternoon)
  Interventions: Other: cardiac coherence

INTERVENTIONS:
Other: cardiac coherence — standard care associated to cardiac coherence training during 3 months

SUMMARY:
ThThe aim of this study is to determinate the potential benefits of a respiratory training program (cardiac coherence, CC) in patients suffering from acute stress disorder, after a potentially traumatic event. Using this method is supposed to prevent the onset of chronic post traumatic stress disorder after 3 months.

This pilot study will help to determinate the need of developing this kind of complementary and alternative program, and will also provide knowledge about the feasibiility and acceptability of this program for the patients.

DETAILED DESCRIPTION:
Each patient will be teached how to use cardiac coherence with a trained practitioner at the inclusion visit. A respiratory guide on smartphone will be given to the patient aswell as a diary in order to keep tracks of the patient's compliance to this program.

ELIGIBILITY:
Inclusion Criteria:

* patients seen at medico-psychological emergency cell
* patients with an acute stress disorder, diagnosed by DSM-5
* patients who have experienced a potentially traumatic event for the last 3-15 days (vctim or witness)
* patients able to read and write in French language
* person affiliated or beneficiary of a social security scheme.
* person who agrees to participate in the study

Exclusion Criteria:

* patients with respiratory pathology not allowing cardiac coherence training
* patients currently practicing a regular respiratory control technique or within the last 6 months
* patients taking beta-blocker, betamimetic, anti-arrhythmic, opioid, antidepressant
* patients with a pacemaker or suffering from severe cardiac illness
* patients with non-stabilized psychiatric disorder at inclusion
* patient taking benzodiazepine unable to wean off in the week following the inclusion
* patients with addiction
* patients with a cognitive deficit
* patients under guardianship or curatorship, under judicial supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients without Post-traumatic stress disorder | at month 3
  Measured by the Post Traumatic Stress Disorder CheckList for DSM-5 (PCL-5)

SECONDARY OUTCOMES:
Complications associated to Post-traumatic stress disorder | at inclusion
  number of suicide attempt
Complications associated to Post-traumatic stress disorder | at month 3
  Variation of suicidal risk (Columbia-Suicide Severity Rating Scale or C-SSRS). This scale measure the risk of suicide et will be measured by un external evaluator
Variation in heart rate variability | at inclusion
  measured by time and frequency indices obtained on the tachogram
Variation in heart rate variability | at month 3
  measured by time and frequency indices obtained on the tachogram
Duration of scale completion | at inclusion
  timed
Duration of scale completion | at month 3
  timed
Compliance to Cardiac coherence | at inclusion
  percentage of time spent in cardiac coherence
Compliance to Cardiac coherence | at month 1
  percentage of time spent in cardiac coherence
Compliance to Cardiac coherence | at month 2
  percentage of time spent in cardiac coherence
Compliance to Cardiac coherence | at month 3
  percentage of time spent in cardiac coherence
Proportion of patients who refuse to participate | up to month 3
  all screened patient will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Erick GOKALSING, Principal Investigator — Etablissement Public de Santé Mentale de La Réunion
Locations (1):
- Etablissement Public de Santé Mentale de La Réunion, Saint-Paul, Reunion

IPD SHARING:
Plan to Share IPD: No